CLINICAL TRIAL: NCT06716177
Title: Clinical Features and Mechanisms of Acute Myocardial Infarction in Patients Without Traditional Cardiovascular Risk Factors
Brief Title: Clinical Features and Linked MEchanisms in Acute Risk-free AMI
Acronym: CLEAR-AMI
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Jiayi Yi, Research Fellow, Beijing Anzhen Hospital
Other Study IDs: KS2024119
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Actue Coronary Syndrome
Keywords: Acute Coronary Syndromes; Risk factor; Multi-omics analysis
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients Without Traditional Cardiovascular Risk Factors Experiencing AMI: This cohort includes patients diagnosed with acute myocardial infarction (AMI) who do not exhibit traditional cardiovascular risk factors such as hypertension, diabetes, dyslipidemia, smoking, or obesity. Participants will undergo comprehensive clinical assessments, including advanced imaging (coronary computed tomography angiography and cardiac magnetic resonance imaging), biomarker profiling, and genetic analyses.
  No direct therapeutic interventions will be applied as part of this study; instead, observational methods will be used to analyze clinical characteristics, identify novel biomarkers, and explore mechanisms contributing to AMI pathogenesis in this population. Data collected from this cohort will provide insights into the unique features and risk profiles of AMI patients without conventional risk factors, potentially informing future diagnostic and therapeutic strategies.

SUMMARY:
This study aims to investigate the clinical characteristics and underlying mechanisms of acute myocardial infarction (AMI) in patients without traditional cardiovascular risk factors, such as hypertension, diabetes, dyslipidemia, or smoking history. By analyzing clinical data, imaging findings, and biomarkers, the research seeks to identify novel risk factors and mechanisms contributing to the pathogenesis of AMI in this unique population. The findings are expected to provide insights into improving diagnostic strategies and developing

DETAILED DESCRIPTION:
Acute myocardial infarction (AMI) is a leading cause of morbidity and mortality worldwide, primarily associated with well-established cardiovascular risk factors such as hypertension, diabetes, dyslipidemia, smoking, and obesity. However, a subset of AMI patients present without these traditional risk factors, posing a diagnostic and therapeutic challenge. This study focuses on the clinical characteristics, pathophysiological mechanisms, and potential novel risk factors associated with AMI in patients who lack conventional cardiovascular risk profiles.

The study will be conducted as a single-center observational analysis involving patients diagnosed with AMI but without a history of hypertension, diabetes, dyslipidemia, smoking, or significant family history of coronary artery disease. Key objectives include:

Characterizing Clinical Features: Analyzing demographic, clinical, and imaging data to identify patterns unique to this patient population.

Identifying Biomarkers: Exploring circulating biomarkers, including inflammatory markers, genetic predispositions, and coagulation abnormalities, that may contribute to AMI development.

Understanding Mechanisms: Investigating potential mechanisms such as microvascular dysfunction, endothelial injury, and autoimmune or hypercoagulable states.

The study will utilize advanced imaging techniques, including coronary computed tomography angiography (CTA) and cardiac magnetic resonance imaging (CMR), to assess coronary anatomy and myocardial tissue characteristics. Genomic and proteomic analyses will be performed to identify genetic and molecular contributors.

By elucidating the clinical and mechanistic profile of AMI in this unique population, the research aims to enhance the understanding of nontraditional pathways leading to AMI. These findings will pave the way for improved diagnostic tools, risk stratification models, and novel therapeutic interventions tailored to this underexplored patient group.

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed with acute myocardial infarction (AMI) based on standard clinical criteria (e.g., troponin elevation, ischemic symptoms, or imaging evidence of myocardial injury).

Absence of traditional cardiovascular risk factors, including hypertension, diabetes, dyslipidemia, smoking, or obesity (BMI < 30 kg/m²).

Aged 18 years or older. Willing and able to provide informed consent.

Exclusion Criteria:

Presence of any traditional cardiovascular risk factors as defined above. History of known congenital or structural heart disease. Severe systemic diseases that could independently contribute to AMI (e.g., severe infection, malignancy, or autoimmune disorders).

Recent history of major surgery or trauma within the last 3 months. Pregnancy or lactation. Inability to provide informed consent due to cognitive impairment or other reasons.

Participation in another interventional clinical trial that might interfere with study outcomes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes patients diagnosed with acute myocardial infarction (AMI) who lack traditional cardiovascular risk factors such as hypertension, diabetes, dyslipidemia, smoking, and obesity. These patients are recruited from a single-center or multicenter setting, such as hospitals with advanced cardiac care facilities.
  The population represents a unique subset of AMI patients, often underexplored in existing research. Comprehensive data, including demographic information, clinical presentations, imaging findings, laboratory biomarkers, and genetic profiles, will be collected to investigate novel risk factors and pathophysiological mechanisms contributing to AMI in this group. The study seeks to provide a detailed understanding of the characteristics and etiology of AMI in this nontraditional population.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Acute Myocardial Infarction (AMI) Without Traditional Cardiovascular Risk Factors | 5 years
  The primary outcome measure is the identification and characterization of acute myocardial infarction (AMI) cases occurring in patients who lack traditional cardiovascular risk factors, such as hypertension, diabetes, dyslipidemia, smoking, or obesity. The outcome will be evaluated by analyzing clinical presentation, laboratory biomarkers, imaging findings, and other diagnostic criteria to confirm the occurrence of AMI and its distinct features in this unique patient population. This will be assessed at the time of diagnosis and through follow-up evaluations during the study period.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shamaki GR, Safiriyu I, Kesiena O, Mbachi C, Anyanwu M, Zahid S, Rai D, Bob-Manuel T, Corteville D, Alweis R, Batchelor WB. Prevalence and Outcomes in STEMI Patients Without Standard Modifiable Cardiovascular Risk Factors: A National Inpatient Sample Analysis. Curr Probl Cardiol. 2022 Nov;47(11):101343. doi: 10.1016/j.cpcardiol.2022.101343. Epub 2022 Aug 5. PMID 35934021
- [Background] Vernon ST, Coffey S, D'Souza M, Chow CK, Kilian J, Hyun K, Shaw JA, Adams M, Roberts-Thomson P, Brieger D, Figtree GA. ST-Segment-Elevation Myocardial Infarction (STEMI) Patients Without Standard Modifiable Cardiovascular Risk Factors-How Common Are They, and What Are Their Outcomes? J Am Heart Assoc. 2019 Nov 5;8(21):e013296. doi: 10.1161/JAHA.119.013296. Epub 2019 Nov 1. PMID 31672080
- [Background] Anderson JL, Knight S, May HT, Le VT, Almajed J, Bair TL, Knowlton KU, Muhlestein JB. Cardiovascular Outcomes of ST-Elevation Myocardial Infarction (STEMI) Patients without Standard Modifiable Risk Factors (SMuRF-Less): The Intermountain Healthcare Experience. J Clin Med. 2022 Dec 22;12(1):75. doi: 10.3390/jcm12010075. PMID 36614876
- [Background] Chandrashekhar Y, Alexander T, Mullasari A, Kumbhani DJ, Alam S, Alexanderson E, Bachani D, Wilhelmus Badenhorst JC, Baliga R, Bax JJ, Bhatt DL, Bossone E, Botelho R, Chakraborthy RN, Chazal RA, Dhaliwal RS, Gamra H, Harikrishnan SP, Jeilan M, Kettles DI, Mehta S, Mohanan PP, Kurt Naber C, Naik N, Ntsekhe M, Otieno HA, Pais P, Pineiro DJ, Prabhakaran D, Reddy KS, Redha M, Roy A, Sharma M, Shor R, Adriaan Snyders F, Weii Chieh Tan J, Valentine CM, Wilson BH, Yusuf S, Narula J. Resource and Infrastructure-Appropriate Management of ST-Segment Elevation Myocardial Infarction in Low- and Middle-Income Countries. Circulation. 2020 Jun 16;141(24):2004-2025. doi: 10.1161/CIRCULATIONAHA.119.041297. Epub 2020 Jun 15. PMID 32539609
- [Background] Roth GA, Mensah GA, Johnson CO, Addolorato G, Ammirati E, Baddour LM, Barengo NC, Beaton AZ, Benjamin EJ, Benziger CP, Bonny A, Brauer M, Brodmann M, Cahill TJ, Carapetis J, Catapano AL, Chugh SS, Cooper LT, Coresh J, Criqui M, DeCleene N, Eagle KA, Emmons-Bell S, Feigin VL, Fernandez-Sola J, Fowkes G, Gakidou E, Grundy SM, He FJ, Howard G, Hu F, Inker L, Karthikeyan G, Kassebaum N, Koroshetz W, Lavie C, Lloyd-Jones D, Lu HS, Mirijello A, Temesgen AM, Mokdad A, Moran AE, Muntner P, Narula J, Neal B, Ntsekhe M, Moraes de Oliveira G, Otto C, Owolabi M, Pratt M, Rajagopalan S, Reitsma M, Ribeiro ALP, Rigotti N, Rodgers A, Sable C, Shakil S, Sliwa-Hahnle K, Stark B, Sundstrom J, Timpel P, Tleyjeh IM, Valgimigli M, Vos T, Whelton PK, Yacoub M, Zuhlke L, Murray C, Fuster V; GBD-NHLBI-JACC Global Burden of Cardiovascular Diseases Writing Group. Global Burden of Cardiovascular Diseases and Risk Factors, 1990-2019: Update From the GBD 2019 Study. J Am Coll Cardiol. 2020 Dec 22;76(25):2982-3021. doi: 10.1016/j.jacc.2020.11.010. PMID 33309175